CLINICAL TRIAL: NCT00236249
Title: Evaluation of Lidocaine Continuous Intravenous Administration for Postoperative Recovery After Colorectal Surgery
Brief Title: Safety and Efficacy Study of Intravenous Lidocaine After Colorectal Surgery: LIDOREHAB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Myriem CARRIER, Department of Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P041008
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2007-03

CONDITIONS: Colorectal Neoplasms
Keywords: Double blind method; Prospective study; Lidocaine/administration and dosage/therapeutic use; Anaesthetics local/administration and dosage; Opioids/administration and dosage; Pain, postoperative; Perioperative care; Postoperative care; Analgesia, Patient-controlled; Length of stay; Survival analysis; Patient satisfaction; Surgery; Middle age; Adult; Aged
MeSH Terms: conditions — Colorectal Neoplasms; Pain, Postoperative; Agnosia; Patient Satisfaction | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lidocaine

SUMMARY:
The purpose of this study is to check if lidocaine intravenous administration during surgery and 24 hours after surgery, associated with standardised management of the patient, helps to accelerate recovery and to improve the quality of recovery, after surgery for colic or rectal neoplasms.

DETAILED DESCRIPTION:
One of the purposes of postoperative care is to shorten the duration of recovery, in order to reduce the complications and to improve the quality of life. After abdominal surgery, two factors can be modified: early mobilisation, thanks to optimal pain control, and return to a normal feeding, permitted by transit recovery. Opioids, which are usually used for pain control, delay the intestinal transit and can be responsible for side effects like drowsiness, nausea, urine retention.

Lidocaine is a local anaesthetic, which means that it can stop the pain if it is administrated around the nerves. It can also be used intravenously. In this way, it is supposed to decrease opioid consumption, accelerate intestinal transit and even decrease inflammation. Side effects of lidocaine appear at higher plasma concentrations than those considered in the study.

After randomisation, the patient will receive either intravenous lidocaine during the surgery and 24 hours after the surgery, or physiological serum (like placebo). Every patient will dispose of patient-controlled-analgesia with morphine and of a standardised care management. Data will be collected concerning pain level, morphine consumption, psychomotor performances, duration of ileus, speed of activity recovery, quality of recovery, and side effects. Biological evaluation of lidocaine concentration and inflammation will also be done.

ELIGIBILITY:
Inclusion Criteria:

* Colorectal neoplasm
* Radical surgery
* Median incision

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) score equal to or up to 3
* Unwilling or unable to use patient-controlled analgesia (PCA)
* Chronic consumption of opioids
* Chronic drug or alcohol abuse
* Chronic pain
* Unable to read or write text
* Inflammatory disease of intestinal tract
* Allergy to morphine
* Allergy to lidocaine
* Severe atrioventricular conduction dysfunction without stimulator
* Porphyry
* Uncontrolled epilepsy
* History of malign hyperthermia
* Severe cardiac failure
* Hepatic failure
* Myasthenia
* Treatment with beta blockers, antiarrhythmic calcium blockers, sultopride, nonselective monoamine oxidase inhibitor (MAOI)
* Locoregional anaesthesia planned
* Associated surgery concerning liver, pancreas, or gall bladder
* Laparoscopic surgery
* Severe psychiatric pathology
* Refusal of the patient

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2005-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Readiness for discharge, checked twice a day

SECONDARY OUTCOMES:
Pain every 4 hours the first day after surgery, then twice a day
Morphine consumption: dose of titration, then twice a day
Time of transit recovery
Physical rehabilitation score daily
Psychomotor test daily until reaching of preoperative values
Quality of recovery score at 1st, 3rd, and 6th day
Satisfaction score at discharge
Biological inflammation the day before the surgery, then at 1st, 3rd, and 6th day
Lidocaine concentration at the end of surgery and 24 hours forward
Clinical side effects twice a day

CONTACTS AND LOCATIONS:
Overall Officials: Claude Jolly, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Saint-Antoine, Paris, France